CLINICAL TRIAL: NCT04995757
Title: Prospective, Randomized, Controlled, Open Label, Single Blinded, All China, Multi-Center, Registration Trial of the Thrombectomy System for the Treatment of Acute Ischemic Stroke.
Brief Title: CAPTURE Registration Trial of the Thrombectomy System for the Treatment of Acute Ischemic Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jian-min Liu, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-GATOR-01-A
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MicroPort NeuroTech Stentretriever (Experimental)
  Interventions: Device: Stent Retriever
- Solitaire FR (Active Comparator)
  Interventions: Device: Stent Retriever

INTERVENTIONS:
Device: Stent Retriever — Stent Retriever for acute ischemic stroke

SUMMARY:
As this will be a pre-market registration trial, in which devices will be used in accordance with appropriately labeled indications, pre-study notifications and approval requests will be addressed with CFDA. All trial results will be shared with CFDA.

ELIGIBILITY:
Inclusion Criteria:

* Subject must demonstrate clinical signs and symptoms that are attributable to the targeted lesion and are consistent with the diagnosis of acute ischemic stroke (AIS), as confirmed by a neuroradiologist (or equivalent expert), using appropriate imaging. Arterial occlusion of ICA, MCA-M1 or MCA-M2.
* Female or male subject, who, at the time of consenting, is aged between 18 and 80 years, inclusive.
* Within 6 hours of stroke symptom onset, subject must have undergone treatment initiation (vascular access through puncture or cut down).
* Signed Informed Consent Form (ICF) completed by subject or subject's legal representative.

Exclusion Criteria:

* 1. Functional dependence prior to stroke onset, defined as a pre-stroke modified Rankin Scale (mRS) score of ≥2.
* 2. Subject's baseline NIHSS score <2 or >25.
* 3. History of severe head injury within past 90 days with residual neurological deficit, as determined by medical history.
* 4. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, e.g. dementia with prescribed anti-cholinesterase inhibitor.
* 5. Seizures at stroke onset if it makes the diagnosis of stroke doubtful and precludes obtaining an accurate baseline NIHSS assessment.
* 6. Subject has a known hemorrhagic diathesis, coagulation factor deficiency; or, is on oral anticoagulant therapy and has an International Normalized Ratio (INR) >3.
* 7. Subject's baseline platelet count is <30*10^9/L.
* 8. Subject's baseline glucose is <50 mg/dL (2.78 mmol/L) or >400 mg/dL (22.2 mmol/L).
* 9. Renal failure, as defined by a serum creatinine >3.0 mg/dL (264 µmol/L) [NOTE: subjects on renal dialysis may be treated regardless of serum creatinine levels].
* 10. Severe, sustained hypertension (SBP > 185 mm Hg or DBP > 110 mmHg) [if the blood pressure can be successfully reduced and maintained at the acceptable level, using medication, the patient can be enrolled].
* 11. Subject has known allergy or contraindication to one or more of the following: anti-platelet drugs; contrast dye; and/or, local or general anesthesia.
* 12. Subject has known allergy to nickel, cobalt chromium, tungsten, platinum or other metal that may be a component of a required medical device needed for treatment.
* 13. Subject is generally unsuitable for endovascular intervention or anesthesia.
* 14. Subject has had major surgery within the previous 30 days
* 15. Subject is an active participant in another drug or device treatment trial for any disease state; or, subject is expected to start participation in another drug or device trial while enrolled in this protocol.
* 16. Subject currently has infective endocarditis or other severe, active bacterial infection.
* 17. Subject's life expectancy is less than 6 months.
* 18. Female of childbearing potential who is known to be pregnant and/or lactating or who has a positive pregnancy test on admission.

Imaging Exclusion Criteria:

* 19. Subject has CT scan or MRI evidence of the following:

  * Significant mass effect with midline shift.
  * Evidence of intracranial tumor, except small meningioma.
  * Evidence of intracranial hemorrhage.
  * Evidence of internal carotid artery flow limiting dissection.
  * Suspected cerebral vasculitis.
  * Suspected aortic dissection.
  * Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation) or clinical evidence of bilateral strokes or strokes in multiple territories.
* 20. The presence of a large completed territorial infarction by non-contrast CT (NCCT), defined as an Alberta Stroke Program Early CT Score (ASPECTS) ≤5.
* 21. Other unusual morphology or lesion that might interfere with device use, including but not limited to the following:

  * Carotid dissection
  * Vasculitis
  * Aortic dissection
  * Aneurysm
  * No transfemoral or alternative access, such as:

    1. Severe intracranial tortuosity
    2. Severe intracranial vasospasm, unresponsive to pharmacotherapy.
    3. Other anatomical or clinical conditions contraindicated for access.
* 22. Anterior circulation strokes involving > 1/3 of the MCA territory, as determined by hypo-density on the baseline non-contrast CT, or low CBV on CT Perfusion imaging, or restricted diffusion on DWI images.
* 23. Thrombotic occlusion in the posterior circulation arteries (vertebral, basilar, etc.)
* 24. Intracranial stent implanted in the same vascular territory that would preclude the safe deployment/removal of the thrombectomy device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-07-05 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Successful Recanalization Rate | immediate post-thrombectomy (t-0) and no later than 3 hours' post-procedure (t-3)
  Defined as modified treatment in cerebral infarction (mTICI) ≥ 2b

SECONDARY OUTCOMES:
mRS at D90 | 90± 14 days' post-treatment
  The modified Rankin Scale (mRS), a combined clinical/functionality and secondary safety endpoint, reflects the degree of disability or dependence in activities of daily living among treated patients. Though listed and classified separately, in multiple publications, as a functionality or clinical endpoint and because of its prominent and unique value in stroke trials, mRS should be considered first among key safety parameters in subjects who complete the 90-day evaluation.
  A successful endpoint will be defined as follows: "at 90± 14 days' post-treatment, the frequency of mRS scores ≤2 or a post-treatment decrease in mRS score of ≥2, relative to the baseline determination". Patients who die, between thrombectomy initiation and 90-Days, will be given an mRS value of 6 in this analysis.
Time from puncture to mTICI≥2b | immediate post-thrombectomy (t-0)
  Time from puncture to mTICI≥2b
The NIHSS score at 30H post-treatment | 30± 6 hours' post-treatment
  The NIHSS score at 30H post-treatment
Symptomatic intracranial hemorrhage(sICH) within 30H post-treatment | 30±6 hours' post-treatment
  Any intracranial hemorrhage judged by CT(or MRI) with neurological symptoms
Death within 90D post-treatment | 90± 14 days' post-treatment
  Any cause death within 90D post-treatment
AE/SAE within 90D post-treatment | 90± 14 days' post-treatment
  Any cause AE/SAEs within 90D post-treatment
Stentretriever/procedure/stroke related AE/SAEs within 90D post-treatment | 90± 14 days' post-treatment
  Stentretriever/procedure/stroke related AE/SAEs within 90D post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai City, China

REFERENCES:
- [Derived] Li G, Sun Y, Liu T, Yang P, Peng Y, Chen W, Zhang L, Chu J, Kuai D, Wang Z, Wu W, Xu Y, Zhou B, Geng Y, Yin C, Li J, Wang M, Peng X, Xiao Y, Li M, Zhang X, Liu P, Wang N, Zhang Y. Predictive factors of poor outcome and mortality among anterior ischaemic stroke patients despite successful recanalisation in China: a secondary analysis of the CAPTURE trial. BMJ Open. 2023 Dec 9;13(12):e078917. doi: 10.1136/bmjopen-2023-078917. PMID 38070920
- [Derived] Zhang Y, Liu P, Li Z, Peng Y, Chen W, Zhang L, Chu J, Kuai D, Chen Z, Wu W, Xu Y, Zhang Y, Zhou B, Geng Y, Yin C, Li J, Wang M, Zhai N, Peng X, Ji Z, Xiao Y, Zhu X, Cai X, Zhang L, Hong B, Xing P, Shen H, Zhang Y, Li M, Shang M, Liu J, Yang P. Endovascular treatment of acute ischemic stroke with a fully radiopaque retriever: A randomized controlled trial. Front Neurol. 2022 Dec 14;13:962987. doi: 10.3389/fneur.2022.962987. eCollection 2022. PMID 36588884